CLINICAL TRIAL: NCT01001312
Title: Treating to Euvolemia by Clinical Assessment and Measured Blood Volume in Heart Failure
Brief Title: Safety and Efficacy of Direct Blood Volume Measurement in the Treatment of Heart Failure
Acronym: TEAM-HF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: NYU Langone Health (Other)
Collaborators: Daxor Corporation (Industry)
Responsible Party: Principal Investigator, Stuart Katz, Principal Investigator, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H09-560
Record Dates: First submitted 2009-10-22; First posted 2009-10-26 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure
Keywords: Heart Failure; Therapeutics; Blood volume
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daxor Blood Volume Analysis (Experimental): Subjects in this treatment arm will receive guideline recommended treatment based on direct blood volume measurement for assessment of volume status.
  Interventions: Other: Daxor Blood Volume Analysis
- Clinical volume status assessment (Active Comparator): Subjects in this treatment arm will receive guideline recommended treatment based on clinical assessment of volume status.
  Interventions: Other: Clinical volume status assessment

INTERVENTIONS:
Other: Daxor Blood Volume Analysis — Radiolabeled albumin for direct measurement of blood volume
  Arms: Daxor Blood Volume Analysis
Other: Clinical volume status assessment — Volume assessment based on history and physical examination
  Arms: Clinical volume status assessment

SUMMARY:
Heart failure is a common cardiac condition affecting nearly 6 million Americans. Silent blood volume overload is common in patients with heart failure and is associated with increased risk of death. This study is designed to determine if adjustment of therapy based on direct measurement of blood volume will reduce risk of hospitalization and death when compared with therapy based on clinical assessment of blood volume in patients with chronic heart failure.

DETAILED DESCRIPTION:
Multicenter prospective randomized trial to compare heart failure management strategies based on clinical assessment of volume status vs. direct measurement of blood volume with a radioisotope technique. Subjects will be randomly assigned to a standard care strategy with guideline recommended treatment based on serial clinical assessment of blood volume or a measured blood volume strategy with guideline recommended treatment based on serial measured blood volume. All subjects will undergo blood volume measurement procedures, but the testing results will only be returned to the physician in the group assigned to management according to measured blood volume status. Subjects will be blinded to their study treatment assignment status.

ELIGIBILITY:
Inclusion Criteria:

* Age >21 years
* Discharge from hospital or emergency department observation unit with a primary diagnosis of acute decompensated heart failure
* Planned discharge home
* Able and willing to provide informed consent

Exclusion Criteria:

* Significant co-morbidity during heart failure hospitalization (treated pneumonia, sepsis, respiratory failure, oliguric renal failure, major bleeding requiring transfusion, stroke)
* Heart failure primarily due to significant valvular disease, sub-aortic outflow obstruction, active myocardial ischemia, apical ballooning syndrome, active arrhythmias, active myocarditis, primary restrictive cardiomyopathy, pericardial disease, or congenital heart disease
* Other major co-morbidities that increase mortality risk (stroke with hemiplegia, diabetes with end-organ damage other than heart disease, history of cancer in last 2 years, moderate to severe liver disease, HIV infection with AIDS)
* Hospitalization length of stay >10 days
* Evidence of acute coronary syndrome during qualifying heart failure hospitalization
* Planned revascularization procedure within 6 months
* Planned implantation of ICD or pacemaker within 6 months
* Planned placement on cardiac transplantation list within 6 months
* Planned other major cardiac surgery or other surgery within 6 months
* Planned intermittent or continuous intravenous positive inotropic therapy
* Planned intermittent or continuous intravenous vasodilator therapy
* Severe obesity (BMI ≥ 40 kg/m2) or cachexia (BMI ≤18 kg/m2)
* Severe chronic kidney disease (estimated GFR<30 ml/min (Modification of Diet in Renal Disease formula20))
* Hemoglobin < 10 gm/dl
* Non-cardiac primary limitation to exercise (rheumatological, orthopedic, pulmonary, neurological or peripheral vascular disease)
* Known history of non-adherence with medications
* Psycho-social factors that interfere with ability to adhere to study procedures (dementia, active substance abuse, poorly controlled psychiatric illnesses, inability to travel frequently to the study center)
* Pregnant women or nursing mothers
* Women of childbearing potential not using adequate birth control methods
* Known hypersensitivity to iodine, eggs, or any other component of the Volumex injection kit
* History of anaphylaxis
* Participation in another heart failure investigational treatment protocol currently or <30 days

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Hospitalization-free Survival | 6 months

SECONDARY OUTCOMES:
Cardiovascular mortality | 6 months
Heart failure hospitalization | 6 months
Quality of life questionnaire (KCCQ) | 6 months
6 minute walk test | 6 months
Hospitalization for worsening renal function | 6 months
All cause hospitalization | 6 months
All cause mortality | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stuart D Katz, M.D., Principal Investigator — NYU School of Medicine
Locations (9):
- United States (9):
  - Pacific Cardiology LLC, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - Baltimore VA Medical Center, Baltimore, Maryland
  - Valley Hospital, Ridgewood, New Jersey
  - New York University Langone Medical Center, New York, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - St. Luke's Regional Heart Center-Bethlehem, Bethlehem, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - St. Thomas Research Institute, Nashvilled, Tennessee